CLINICAL TRIAL: NCT02735239
Title: Phase 1/2 Study of Anti-PD-L1 in Combination With Chemo(Radio)Therapy for Oesophageal Cancer
Brief Title: Study of Anti-PD-L1 in Combination With Chemo(Radio)Therapy for Oesophageal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUD2015-005; 2015-005298-19 (EudraCT Number); ESR 15-10891 (Other: AstraZeneca reference number)
Record Dates: First submitted 2016-03-17; First posted 2016-04-12 (Estimated); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-09

CONDITIONS: Esophageal Cancer
Keywords: Oesophageal Cancer; Oesophageal adenocarcinoma; Oesophageal squamous cell carcinoma; Immunotherapy; Cytotoxic T-lymphocyte-associated protein 4 (CTLA-4); Programmed cell death protein 1 (PD-1); Programmed death ligand 1 (PD-L1)
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Diabetes Mellitus, Insulin-Dependent, 12; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — durvalumab; tremelimumab; Oxaliplatin; Capecitabine; Radiotherapy; Radiation; Paclitaxel; Carboplatin; Fluorouracil; Leucovorin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort A1: Metastatic/locally advanced OC, Durva + Chemotherapy (Chemo) (Experimental): Durvalumab (750 mg IV every two weeks [Q2W]) was to be given for up to 11 doses. Oxaliplatin (130 mg/m^2 IV)/capecitabine (1250 mg/m^2/day given orally) chemotherapy was started on the day of the third dose of durvalumab and continued for 6 doses.
  Interventions: Drug: Durvalumab; Drug: Oxaliplatin; Drug: Capecitabine
- Cohort A2: Metastatic/locally advanced OC, Durva, Treme + Chemo (Experimental): Durvalumab (750 mg IV Q2W) was to be given for up to 11 doses. One dose of tremelimumab (37.5 mg IV) was given on the same day as the first dose of durvalumab. Oxaliplatin (130 mg/m^2 IV)/capecitabine (1250 mg/m^2/day given orally) chemotherapy was started on the day of the third dose of durvalumab and continued for 6 doses.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Oxaliplatin; Drug: Capecitabine
- Cohort B: Metastatic/locally advanced OC, Durva, Treme + Chemo (Experimental): Durvalumab (750 mg IV Q2W) was to be given for up to 11 doses. One dose of tremelimumab (75 mg IV) was given on the same day as the first dose of durvalumab. Oxaliplatin (130 mg/m^2 IV)/capecitabine (1250 mg/m^2/day given orally) chemotherapy was started on the day of the third dose of durvalumab and continued for 6 doses.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Oxaliplatin; Drug: Capecitabine
- Cohort C: Operable OC; Durva + Chemo (Experimental): Durvalumab (750 mg IV Q2W) was to be given for up to 5 doses. Two cycles of neoadjuvant oxaliplatin (130 mg/m^2 IV)/capecitabine (1250 mg/m^2/day given orally) chemotherapy were to be administered before surgery. Subjects were to undergo surgery 6 to 8 weeks after completing chemotherapy or according to institutional policies for surgery; and would be eligible to resume durvalumab dosing (to a maximum of 12 infusions) once recovered from surgery, provided that this was within 3 months of surgery.
  Interventions: Drug: Durvalumab; Drug: Oxaliplatin; Drug: Capecitabine
- Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy (Experimental): Durvalumab (750 mg IV Q2W) was to be given for up to 6 doses. Two cycles of neoadjuvant 5-fluorouracil (5-FU) (2600 mg/m^2 24-hr IV), leucovorin (200 mg/m^2 IV), oxaliplatin (85 mg/m^2 IV), and docetaxel (50 mg/m^2 IV) chemotherapy (FLOT) were to be administered before surgery starting on the day of the third dose of durvalumab. Subjects were to undergo surgery 6 to 8 weeks after completing chemotherapy or according to institutional policies for surgery; and would be eligible to resume durvalumab dosing (to a maximum of 12 infusions), FLOT or durvalumab plus FLOT at the discretion of the Investigator once recovered from surgery, provided that this was within 3 months of surgery.
  Interventions: Drug: Durvalumab; Drug: Oxaliplatin; Drug: 5-fluorouracil (5-FU); Drug: Leucovorin; Drug: Docetaxel
- Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(radio)therapy (Experimental): Durvalumab (750 mg IV Q2W) was to be given for 2 doses. This was followed by five weekly doses of neoadjuvant paclitaxel (50 mg/m^2 IV) / carboplatin (AUC 2) IV chemotherapy + radiotherapy (41.4 Gy radiotherapy given over 23 fractions) before surgery. Subjects could receive an additional dose of durvalumab after completion of chemoradiation.
  In Cohort D2, subjects continued durvalumab for 3 additional doses while receiving chemoradiation. Subjects were to undergo surgery 6 to 8 weeks after completing chemo(radio)therapy or according to institutional policies for surgery; and would be eligible to resume durvalumab dosing (to a maximum of 12 infusions) once recovered from surgery, provided that this was within 3 months of surgery.
  Interventions: Drug: Durvalumab; Radiation: Radiotherapy; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Durvalumab — Anti PD-L1 antibody
  Other Names: MEDI4736; Imfinzi®; Durva
Drug: Tremelimumab — Anti CTLA-4 antibody
  Other Names: Treme
  Arms: Cohort A2: Metastatic/locally advanced OC, Durva, Treme + Chemo; Cohort B: Metastatic/locally advanced OC, Durva, Treme + Chemo
Drug: Oxaliplatin — IV administered chemotherapy
  Other Names: Eloxatin®
  Arms: Cohort A1: Metastatic/locally advanced OC, Durva + Chemotherapy (Chemo); Cohort A2: Metastatic/locally advanced OC, Durva, Treme + Chemo; Cohort B: Metastatic/locally advanced OC, Durva, Treme + Chemo; Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy; Cohort C: Operable OC; Durva + Chemo
Drug: Capecitabine — orally-administered chemotherapy
  Other Names: Xeloda®
  Arms: Cohort A1: Metastatic/locally advanced OC, Durva + Chemotherapy (Chemo); Cohort A2: Metastatic/locally advanced OC, Durva, Treme + Chemo; Cohort B: Metastatic/locally advanced OC, Durva, Treme + Chemo; Cohort C: Operable OC; Durva + Chemo
Radiation: Radiotherapy
  Other Names: Radiation
  Arms: Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(radio)therapy
Drug: Paclitaxel — IV administered chemotherapy
  Other Names: Taxol®
  Arms: Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(radio)therapy
Drug: Carboplatin — IV administered Chemotherapy
  Other Names: Paraplatin®
  Arms: Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(radio)therapy
Drug: 5-fluorouracil (5-FU) — IV administered chemotherapy
  Other Names: Adrucil®
  Arms: Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy
Drug: Leucovorin — chemo-protective agent
  Other Names: Leucovorin calcium; Folinic Acid
  Arms: Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy
Drug: Docetaxel — IV administered chemotherapy
  Other Names: Taxotere®
  Arms: Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy

SUMMARY:
This is an open-label, Phase 1/2 study to evaluate the safety of durvalumab (MEDI4736) in combination with oxaliplatin/capecitabine chemotherapy in metastatic/locally advanced oesophageal cancer (OC) and with neoadjuvant chemo(radio)therapy before surgery in operable OC. The immunotherapy will be given for a 4-week period before starting the standard chemo(radio)therapy, continuing durvalumab treatment once the chemotherapy starts. The study will include 2 phases, a safety run-in Phase 1 (Cohorts A1 and A2) and an expansion Phase 2 (Cohorts B, C, C-FLOT, D/D2).

DETAILED DESCRIPTION:
This is an open-label, Phase 1/2 study to evaluate the safety of immunotherapy in combination with chemo (radio) therapy with the following cohorts:

* Cohorts A1, A2, and B: Oxaliplatin/capecitabine chemotherapy in metastatic/locally advanced oesophageal cancer (OC).
* Cohort C: Neoadjuvant oxaliplatin/capecitabine chemotherapy before surgery in operable OC.
* Cohort C-FLOT: Neoadjuvant 5-fluorouracil (5-FU), leucovorin, oxaliplatin, and docetaxel (FLOT) chemotherapy before surgery in operable OC.
* Cohort D/D2: Neoadjuvant paclitaxel/carboplatin chemotherapy + radiotherapy before surgery in operable OC.

The immunotherapy will be given for a 4-week period before starting the standard chemo(radio)therapy, continuing durvalumab treatment once the chemotherapy starts for all cohorts except Cohort D.

The study will include 2 phases, a safety run-in Phase 1 (Cohorts A1 and A2) and an expansion Phase 2 (Cohorts B including the higher dose tremelimumab cohort from Cohort A2, C, C-FLOT, and D/D2).

Phase 1 will evaluate the safety of durvalumab alone (Cohort A1) administered before chemotherapy (oxaliplatin + capecitabine) in subjects with metastatic or locally advanced OC. After completion of Cohort A1, Phase 2 in Cohorts C, C-FLOT, and D/D2 will begin, and a safety review will determine whether to explore the tremelimumab + durvalumab combination (Cohort A2).

Phase 2 includes the expansion into Cohorts B, C, C-FLOT, and D/D2. Once Cohort A1 is cleared, there will be concurrent enrollment into Phase 2 expansion for Cohorts C, C-FLOT and D/D2 (subjects with operable OC with neoadjuvant chemotherapy or chemoradiotherapy before surgery) and the tremelimumab dose-escalation phase for Cohort A2 (37.5 mg and 75 mg). Once Cohort A2 is completed, another safety review will determine the dose of tremelimumab to be included in the recommended combination dose (RCD) to start enrollment into the Cohort B (subjects with metastatic/locally advanced OC) expansion phase. Subjects treated at the RCD in Cohort A2 (tremelimumab 75 mg) will be included in Cohort B.

Subjects in Cohorts C, C-FLOT and D/D2 will undergo surgery after completing treatment, and they will be eligible to resume durvalumab dosing (to a maximum of 12 infusions) once recovered from surgery, provided that this is within 3 months of surgery. Subjects in Cohort C-FLOT may receive durvalumab, FLOT, or durvalumab plus FLOT at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of oesophageal or gastrooesophageal cancer and have not received prior chemotherapy.

   * Cohorts A and B - metastatic/locally advanced cancer
   * Cohorts C/C-FLOT and D/D2 - deemed suitable for surgery with curative intent
2. Anticipated lifespan greater than 4 months.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. At the time of day 1 of the study, subjects with brain metastases must be asymptomatic for at least 4 weeks and:

   * at least 8 weeks without tumour progression after any whole brain radiotherapy
   * at least 4 weeks since craniotomy and resection or stereotactic radiosurgery
   * at least 3 weeks without new brain metastases as evidenced by MRI/CT
5. Adequate normal organ and marrow function. Laboratory parameters for vital functions should be in the normal range. Laboratory abnormalities that are not clinically significant are generally permitted.
6. Written informed consent obtained from the subject; subject been informed of other treatment options, and able to comply with study requirements.
7. Age 18 years or older.

Exclusion Criteria

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site). Previous enrollment in the present study.
2. Participation in another clinical study with an investigational product during the last 4 weeks.
3. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's Correction.
4. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
5. History of allogeneic organ transplant.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C, known immunodeficiency or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
7. Known history of previous clinical diagnosis of tuberculosis.
8. History of pneumonitis or interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-06-24 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Middleton, Study Chair — University of Oxford, UK
Locations (4):
- United Kingdom (4):
  - Research Facility, Dundee
  - Research Facility, Nottingham
  - Research Facility, Oxford
  - Research Facility, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bohnsack O, Hoos A, Ludajic K. Adaptation of the immune related response criteria: irRECIST. Ann Oncol. 2014 Sep;25(suppl 4):iv361-iv72 [Abstract 4958]. doi: 10.1093/annonc/mdu342.23.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(Radio)Therapy: Durvalumab (750 mg IV Q2W) was to be given for 2 doses. This was followed by five weekly doses of neoadjuvant paclitaxel (50 mg/m^2 IV) / carboplatin (AUC 2) IV chemotherapy + radiotherapy (41.4 Gy radiotherapy given over 23 fractions) before surgery. Subjects could receive an additional dose of durvalumab after completion of chemoradiation.
  In Cohort D2, subjects continued durvalumab for 3 additional doses while receiving chemoradiation. Subjects were to undergo surgery 6 to 8 weeks after completing chemo(radio)therapy or according to institutional policies for surgery; and would be eligible to resume durvalumab dosing (to a maximum of 12 infusions) once recovered from surgery, provided that this was within 3 months of surgery.
  Durvalumab: Anti PD-L1 antibody
  Radiotherapy
  Paclitaxel: IV administered chemotherapy
  Carboplatin: IV administered chemotherapy
Period: Overall Study
Arm/Group | Cohort A1: Metastatic/Locally Advanced OC, Durva + Chemotherapy (Chemo) | Cohort A2: Metastatic/Locally Advanced OC, Durva, Treme + Chemo | Cohort B: Metastatic/Locally Advanced OC, Durva, Treme + Chemo | Cohort C: Operable OC; Durva + Chemo | Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy | Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(Radio)Therapy
Started (All Subjects who received at least one dose of study treatment.) | 12 | 5 | 21 | 11 | 9 | 15
Completed (All subjects who completed protocol specified treatment. For Cohorts C and D/D2 this includes subjects who completed pre-surgery treatment.) | 8 | 2 | 13 | 11 | 9 | 13
Not Completed | 4 | 3 | 8 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Progressive disease | 3 | 1 | 3 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A1: Metastatic/Locally Advanced OC, Durva + Chemotherapy (Chemo) | Cohort A2: Metastatic/Locally Advanced OC, Durva, Treme + Chemo | Cohort B: Metastatic/Locally Advanced OC, Durva, Treme + Chemo | Cohort C: Operable OC; Durva + Chemo | Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy | Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(Radio)Therapy | Total
Number analyzed (Participants) | 12 | 5 | 21 | 11 | 9 | 15 | 73
Age, Continuous [Median (Full Range); unit: years] | 59.5 [23 to 75] | 55.0 [29 to 67] | 58.0 [42 to 78] | 57 [46 to 71] | 56 [33 to 72] | 65 [50 to 72] | 59 [23 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 0 | 1 | 3 | 11
  Male | 10 | 4 | 17 | 11 | 8 | 12 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 12 | 5 | 20 | 11 | 8 | 14 | 70
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12 | 5 | 21 | 11 | 9 | 15 | 73

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Treatment Emergent Adverse Events (TEAEs)
Description: Toxicity was graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. Adverse events (AEs) were reported based on clinical laboratory tests, vital signs, physical examinations, and any other medically indicated assessments, including subject interviews, from the time informed consent is signed through 110 days after the last dose of study treatment. Treatment-emergent AEs were those that occurred or worsened after administration of the first dose of study treatment.
  In Cohorts A1, A2 and B, 12, 5 and 7 subjects, respectively, were monitored for dose limiting toxicities (DLTs) during the first 10 weeks of treatment (DLT evaluation period).
Time Frame: up to 1 year
Population: All subjects who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: Metastatic/Locally Advanced OC, Durva + Chemotherapy (Chemo) | Cohort A2: Metastatic/Locally Advanced OC, Durva, Treme + Chemo | Cohort B: Metastatic/Locally Advanced OC, Durva, Treme + Chemo | Cohort C: Operable OC; Durva + Chemo | Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy | Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(Radio)Therapy
Number analyzed (Participants) | 12 | 5 | 21 | 11 | 9 | 15
Participants
  Treatment-emergent adverse events (TEAEs) | 12 | 5 | 21 | 11 | 9 | 15
  Dose-limiting toxicities (DLTs) during the entire study | 0 | 1 | 2 | 0 | 0 | 0
  Discontinued due to a TEAE | 0 | 0 | 4 | 0 | 0 | 0
  DLTs within the 10-week DLT evaluation period: number analyzed (Participants) | 12 | 5 | 7 | 0 | 0 | 0
  DLTs within the 10-week DLT evaluation period | 0 | 0 | 0 |  |  |

2. Primary Outcome: Number of Subjects With Best Overall Tumor Response by the Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST)
Description: Tumor responses were evaluated using appropriate imaging and categorized according to irRECIST at Screening (up to 28 days before the first dose of study treatment), and in Cycles 1, 3, 5 and 6 in Cohorts A1, A2 and B. In the other cohorts, tumor response was assessed at baseline, post-surgery and 14 days after the last dose. In Cohorts C-FLOT and D, an additional assessment was done prior to surgery and in Cohorts C and D, an additional assessment was done in Cycle 3. Per irRECIST, measurable lesions are categorized as follows: Immune-related Complete Response (irCR): Complete disappearance of all target lesions; Immune-related Partial Response (irPR): ≥ 30% decrease from baseline in the Total Measurable Tumor Burden (TMTB); Immune-related Progressive Disease (irPD): ≥ 20% increase from nadir in TMTB; Immune-related Stable Disease (irSD): not meeting above criteria; irNon-CR/Non-PD: irNon-CR/Non-PD is preferred over SD when no lesions can be measured.
Time Frame: up to 1 year
Population: All subjects who received at least one dose of study treatment and had a baseline and at least one post-baseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: Metastatic/Locally Advanced OC, Durva + Chemotherapy (Chemo) | Cohort A2: Metastatic/Locally Advanced OC, Durva, Treme + Chemo | Cohort B: Metastatic/Locally Advanced OC, Durva, Treme + Chemo | Cohort C: Operable OC; Durva + Chemo | Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy | Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(Radio)Therapy
Number analyzed (Participants) | 11 | 5 | 20 | 9 | 5 | 8
Participants
  irCR | 2 | 0 | 0 | 3 | 1 | 2
  irPR | 3 | 3 | 10 | 1 | 0 | 0
  irSD | 5 | 1 | 4 | 0 | 0 | 0
  irPD | 1 | 1 | 5 | 1 | 0 | 1
  irNon-CR/Non-PD | 0 | 0 | 1 | 1 | 0 | 0
  Not Evaluable | 0 | 0 | 0 | 3 | 4 | 5

3. Secondary Outcome: Number of Subjects With Metastatic/Locally Advanced Oesophageal Cancer (OC) Who Had a Response at Cycle 6 by the Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST)
Description: Tumor responses were evaluated using appropriate imaging and categorized according to irRECIST at Screening (up to 28 days before the first dose of study treatment), and in Cycles 1, 3, 5 and 6 in Cohorts A1, A2 and B. Per irRECIST, measurable lesions are categorized as follows: irCR: Complete disappearance of all target lesions; irPR: ≥ 30% decrease from baseline in the Total Measurable Tumor Burden (TMTB); irPD: ≥ 20% increase from nadir in TMTB; irSD: not meeting above criteria; irNon-CR/Non-PD: irNon-CR/Non-PD is preferred over SD when no lesions can be measured.
Time Frame: Up to 23 weeks
Population: All subjects in Cohorts A1, A2 and B who received at least one dose of study treatment and had a baseline and at least one post-baseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: Metastatic/Locally Advanced OC, Durva + Chemotherapy (Chemo) | Cohort A2: Metastatic/Locally Advanced OC, Durva, Treme + Chemo | Cohort B: Metastatic/Locally Advanced OC, Durva, Treme + Chemo
Number analyzed (Participants) | 8 | 3 | 14
Participants
  irCR | 2 | 0 | 0
  irPR | 2 | 2 | 7
  irSD | 3 | 1 | 4
  irPD | 1 | 0 | 1
  irNon-CR/Non-PD | 0 | 0 | 1
  Not evaluable | 0 | 0 | 1

4. Secondary Outcome: Median Progression-free Survival (PFS) by the Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) as Estimated Using the Kaplan-Meier Method
Description: Tumor responses were evaluated using appropriate imaging and categorized according to irRECIST at Screening (up to 28 days before the first dose of study treatment), and in Cycles 1, 3, 5 and 6 in Cohorts A1, A2 and B. In the other cohorts, tumor response was assessed at baseline, post-surgery and 14 days after the last dose. In Cohorts C-FLOT and D, an additional assessment was done prior to surgery and in Cohorts C and D, an additional assessment was done in Cycle 3.
  In Cohorts A1, A2 and B, PFS was measured from the date of the first dose of study treatment to the date of earliest disease progression according to irRECIST or to the date of death, if disease progression did not occur. For Cohorts C, C-FLOT and D/D2, PFS is measured from the date of surgery. Per irRECIST, irPD was defined as a ≥ 20% increase from nadir in the TMTB.
Time Frame: Up to 3 years
Population: All subjects who received at least one dose of study treatment and had a baseline and at least one post-baseline disease assessment. One subject in Cohort D progressed prior to surgery and as a result was not included in the PFS after surgery assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A1: Metastatic/Locally Advanced OC, Durva + Chemotherapy (Chemo) | Cohort A2: Metastatic/Locally Advanced OC, Durva, Treme + Chemo | Cohort B: Metastatic/Locally Advanced OC, Durva, Treme + Chemo | Cohort C: Operable OC; Durva + Chemo | Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy | Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(Radio)Therapy
Number analyzed (Participants) | 12 | 5 | 21 | 11 | 9 | 14
months | 8.7 [0.9 to 29.1] | 5.2 [1.4 to NA] — Upper limit of the confidence interval not reached due to small number of subjects. | 11.9 [3.9 to 15.6] | 25.4 [6.47 to NA] — Upper limit of the confidence interval not reached due to small number of subjects. | 32.03 [2.10 to NA] — Upper limit of the confidence interval not reached due to small number of subjects. | 9.59 [NA to NA] — Upper and lower limits of the confidence interval not reached due to small number of subjects.

5. Secondary Outcome: Median Overall Survival (OS) as Estimated Using the Kaplan-Meier Method
Description: After completion of treatment, all subjects were followed for survival every 6 months for up to 3 years from start of treatment. OS was measured from the date of the first dose of study treatment to the date of death or last follow-up. Subjects lost to follow-up were censored on the date when they were last known to be alive. Per protocol amendment 8.0, all post study follow-up for the collection of survival data was discontinued as of June 30, 2022.
Time Frame: Up to 3 years
Population: All subjects who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A1: Metastatic/Locally Advanced OC, Durva + Chemotherapy (Chemo) | Cohort A2: Metastatic/Locally Advanced OC, Durva, Treme + Chemo | Cohort B: Metastatic/Locally Advanced OC, Durva, Treme + Chemo | Cohort C: Operable OC; Durva + Chemo | Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy | Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(Radio)Therapy
Number analyzed (Participants) | 12 | 5 | 21 | 11 | 9 | 15
months | 11.8 [3.1 to NA] — Upper limit of the confidence interval not reached due to small number of subjects. | 8.6 [2.7 to NA] — Upper limit of the confidence interval not reached due to small number of subjects. | 15.6 [9.3 to 33.5] | NA [18.46 to NA] — Median and upper limit of the confidence interval not reached due to small number of subjects. | NA [8.02 to NA] — Median and upper limit of the confidence interval not reached due to small number of subjects. | NA [13.14 to NA] — Median and upper limit of the confidence interval not reached due to small number of subjects.

6. Secondary Outcome: One Year Survival Rate in Subjects With Operable OC
Description: OS was measured from the date of the first dose of study treatment to the date of death or last follow-up. Subjects lost to follow-up were censored on the date when they were last known to be alive. Per protocol amendment 8.0, all post study follow-up for the collection of survival data was discontinued as of June 30, 2022.
Time Frame: up to 12 months
Population: All subjects with Operable OC in Cohorts C, C-FLOT and D/D2 who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Cohort C: Operable OC; Durva + Chemo | Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy | Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(Radio)Therapy
Number analyzed (Participants) | 11 | 9 | 15
percent of participants | 100 [NA to NA] — Upper and lower limits of the confidence interval not reached due to small number of subjects. | 89 [43.3 to 98.4] | 86.7 [56.4 to 96.5]

7. Secondary Outcome: Overall Response Prior to Surgery in Operable OC (Cohorts C, C-FLOT and D/D2) Using Positron Emission Tomography (PET) Response Criteria in Solid Tumors (PERCIST)
Description: 18F- fluorodeoxyglucose (18F-FDG) PET scans were conducted at baseline and in Cycle 3 in Cohorts C and D, and after completion of therapy in Cohort C-FLOT and D2. Complete metabolic response: 18F-FDG-avid lesions revert to background of normal tissues in which they are located; Partial metabolic response: 30% or greater reduction in measurable tumors; Stable Metabolic Response: no visible change in metabolic activity of tumor; Progressive metabolic disease: increase in intensity or extent of tumor metabolic activity or new sites of activity.
Time Frame: Up to 7months
Population: All operable OC subjects in Cohorts C, C-FLOT and D/D2 who had a baseline PET scan and a PET scan prior to surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort C: Operable OC; Durva + Chemo | Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy | Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(Radio)Therapy
Number analyzed (Participants) | 11 | 6 | 13
Participants
  Complete Metabolic Response | 2 | 1 | 3
  Partial Metabolic Response | 5 | 3 | 7
  Stable Disease | 1 | 2 | 1
  Progressive Disease | 3 | 0 | 2

ADVERSE EVENTS:
Time Frame: All AEs occurring between the signing of informed consent and the off-study date (i.e., through 110 days after the last dose of study treatment, up 18 months) were documented, regardless of a causal relationship to study drug. AEs that occur or worsen in severity after the first dose of study treatment were considered treatment emergent (i.e., TEAEs). All cause mortality included all deaths which were reported up to 3 years.
Description: AE documentation included onset/resolution dates, severity using NCI CTCAE (version 4.03), seriousness, relationship to study drug, study drug action taken, treatment and outcome. Preferred terms were counted once per subject at the maximum reported grade.
Arm/Group | Cohort A1: Metastatic/Locally Advanced OC, Durva + Chemotherapy (Chemo) | Cohort A2: Metastatic/Locally Advanced OC, Durva, Treme + Chemo | Cohort B: Metastatic/Locally Advanced OC, Durva, Treme + Chemo | Cohort C: Operable OC; Durva + Chemo | Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy | Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(Radio)Therapy
All-Cause Mortality (participants affected / at risk) | 9/12 | 5/5 | 16/21 | 5/11 | 2/9 | 6/15
Serious Adverse Events (participants affected / at risk) | 7/12 | 4/5 | 12/21 | 7/11 | 6/9 | 10/15
Other Adverse Events (participants affected / at risk) | 12/12 | 5/5 | 21/21 | 11/11 | 9/9 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A1: Metastatic/Locally Advanced OC, Durva + Chemotherapy (Chemo) (N=12) | Cohort A2: Metastatic/Locally Advanced OC, Durva, Treme + Chemo (N=5) | Cohort B: Metastatic/Locally Advanced OC, Durva, Treme + Chemo (N=21) | Cohort C: Operable OC; Durva + Chemo (N=11) | Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy (N=9) | Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(Radio)Therapy (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 2 | 1 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 4 | 0 | 0 | 0
Encephalitis autoimmune (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oesophagectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Jejunostomy refashioning (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A1: Metastatic/Locally Advanced OC, Durva + Chemotherapy (Chemo) (N=12) | Cohort A2: Metastatic/Locally Advanced OC, Durva, Treme + Chemo (N=5) | Cohort B: Metastatic/Locally Advanced OC, Durva, Treme + Chemo (N=21) | Cohort C: Operable OC; Durva + Chemo (N=11) | Cohort C-FLOT: Operable OC, Durva + FLOT Chemotherapy (N=9) | Cohort D/D2: Operable OC, Durva + Neoadjuvant Chemo(Radio)Therapy (N=15)
Anaemia (Blood and lymphatic system disorders) | 5 | 1 | 4 | 0 | 3 | 5
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 3 | 0 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1 | 3 | 0 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 1 | 1 | 1
Hypothyroidism (Endocrine disorders) | 2 | 1 | 0 | 1 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 2 | 0 | 2 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 0 | 1
Abdominal distention (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 3 | 1 | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 1 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 4 | 5 | 1 | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 7 | 2 | 11 | 5 | 7 | 10
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 3 | 3 | 4 | 1 | 3 | 3
Epigastric discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 4 | 3 | 3
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 10 | 4 | 12 | 5 | 5 | 9
Lip pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 5
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 11 | 2 | 8 | 1 | 3 | 6
Steatorrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 1 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 3 | 0 | 1 | 2
Early satiety (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 10 | 5 | 13 | 7 | 6 | 8
Influenza like illness (General disorders) | 0 | 1 | 2 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 2 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Infusion site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 0 | 0 | 2 | 0
Temperature intolerance (General disorders) | 0 | 0 | 2 | 3 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Balanitis candida (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 4 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 3 | 0 | 1 | 1 | 2 | 2
Medical device site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Dumping syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 4 | 0 | 1 | 1
Amylase increased (Investigations) | 3 | 1 | 2 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 5 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 2 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 6 | 0 | 1 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 2 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 3 | 4 | 2 | 0 | 4
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 3 | 2 | 5 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 2 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 2 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 2 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 2
Dysaesthesia (Nervous system disorders) | 1 | 0 | 3 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 4 | 0 | 0 | 2 | 3 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Encephalitis autoimmune (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 1 | 1 | 2
Muscle contractions involuntary (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 2 | 6 | 6 | 4 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 3 | 1 | 3 | 3 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 1 | 5 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0
Poor quality sleep (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 2 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 1 | 1 | 0 | 0 | 2
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 4 | 6 | 2 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 3 | 1 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 2
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 5 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 2 | 1 | 2
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0 | 4 | 5
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT02735239/Prot_SAP_000.pdf